CLINICAL TRIAL: NCT03300661
Title: Open-label, Non-Pharmacological, Intervention Cohort Study Without Control Arm, in Patients With Non Alcoholic Fatty Liver Disease and in Healthy Subjects.
Brief Title: Non Alcoholic Fatty Liver Disease: Nutritional Epidemiology and Lifestyle Medicine
Acronym: SEELN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Chiara Ricci, Associate Professor, Università degli Studi di Brescia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ubrescia
Record Dates: First submitted 2017-09-28; First posted 2017-10-03 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Non Alcoholic Fatty Liver Disease; Lifestyle; Diet Modification
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: A single cohort of patients with NAFLD, without control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mediterranean Style (Experimental): Educational intervention with personalized suggestions to improve diet and physical activity
  Interventions: Behavioral: Mediterranean Style

INTERVENTIONS:
Behavioral: Mediterranean Style — After completion of a Food Frequency Questinnaire (FFQ) and the International Physical Activity Questionnaire (IPAQ), patients enrolled in the study undergo a personalized educational intervention by a registered dietician. During the intervention the dietician advice about the main errors in diet and physical activity (by FFQ and IPAQ) and chooses three aims in diet modification and one aim in physical activity improvement. Patients adherence is assessed by the same dietician every three months, using FFQ and IPAQ, and futher supports are provided. Total intervention lenght is twelve months.

SUMMARY:
The study is an open-label intervention non pharmacological Cohort Study without control arm in patients with Non Alcoholic Fatty Liver Disease (NAFLD) and in healthy subjects.

The intervention in patients with NAFLD is educational, providing personalized suggestions to improve diet and physical activity; the intervention in healthy subjects is educational, providing general suggestions to improve diet and physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Presence of Fatty Liver at ultrasonography

Exclusion Criteria:

* Pregnancy;
* Breast Feeding
* Cirrhosis or End Stage Liver Disease
* Fatty Liver due to Hepatic Diseases other than Non Alcoholic Fatty Liver disease
* Concomitant severe clinical condition

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
Weight loss | 12 months
  A reduction of at least 3 Kg
Body Mass Index (BMI) decrease | 12 months
  A dicresae of at least 1Kg/m2
Waist Circumference (WC) decrease | 12 months
  A decrease of at least 1.5 cm

SECONDARY OUTCOMES:
Blood sugar level decrease | 12 months
  A decrease of 6 mg/dL
Blood cholesterol level decrease | 12 months
  A decrease of 9 mg/dL
Blood triglycerides level dicrease | 12 months
  A decrease of 12 mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Ricci, MD. PhD, Principal Investigator — Università degli Studi di Brescia
Locations (1):
- ASST Spedali Civili Brescia, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zanini B, Benini F, Marullo M, Simonetto A, Rossi A, Cavagnoli P, Bonalumi A, Marconi S, Pigozzi MG, Gilioli G, Valerio A, Donato F, Castellano M, Ricci C. Mediterranean-Oriented Dietary Intervention Is Effective to Reduce Liver Steatosis in Patients with Nonalcoholic Fatty Liver Disease: Results from an Italian Clinical Trial. Int J Clin Pract. 2024 Jan 25;2024:8861126. doi: 10.1155/2024/8861126. eCollection 2024. PMID 38303926